CLINICAL TRIAL: NCT00302627
Title: Pamidronate, Vitamin D, and Calcium for the Bone Disease of Kidney and Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: The Heart Institute of Spokane (Unknown); Ochsner Health System (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HI497
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Transplant Bone Disease
Keywords: bisphosphonates; vitamin D; calcium supplement; corticosteroid therapy; fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Pamidronate; Vitamin D; Transplantation; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pamidronate, Vitamin D, and Calcium (Experimental): 60mg or 90mg given at baseline, 6,12,18, and 24 months
  vitamin D 800 units/day
  calcium carbonate 1500 milligrams/day
  Interventions: Drug: Pamidronate; Drug: vitamin D; Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Pamidronate — 60mg or 90mg given at baseline, 6,12,18, and 24 months
  Other Names: Transplant Bone Disease
Drug: vitamin D — baseline, 6,12 months
  Other Names: Vitamin D administration in Transplant
Drug: Calcium Carbonate — baseline, 6,12 months
  Other Names: Calcium administration in Transplant

SUMMARY:
Bone is lost rapidly and fractures occur in 10-20% of patients who receive organ transplants within 2 years. The purpose of this study is to evaluate long-term effects of a pamidronate-vitamin D-calcium regimen on bone loss, fractures, and safety in recipients of kidney and heart transplants.

DETAILED DESCRIPTION:
Pamidronate improves bone mass in numerous disorders of bone. Other bisphosphonates, as well as pamidronate, have been proven to be beneficial in steroid-related bone disorders. Steroid treatment is a major cause of bone loss after organ transplantation. Small, short-term studies suggest that pamidronate prevents bone loss in kidney and heart transplant recipients.

Many bisphosphonates cannot be used in patients with decreased kidney function. However, pamidronate can be given to these patients. This is an advantage of pamidronate in kidney and heart transplantation because of the frequent occurrence of decreased kidney function in these groups. Another advantage of pamidronate is that it is administered intravenously. Oral bisphosphonates commonly produce esophagitis, which is a challenging problem in the transplant population. Potential side-effects of pamidronate include transient hypocalcemia, lymphopenia, low-grade fever, myalgias and nausea. Recently, rare cases of proteinuria and kidney failure were reported in cancer patients receiving high-dose pamidronate. Although this side effect has not been reported in other types of patients receiving pamidronate, this is a safety concern that warrants further scrutiny in the transplant population.

In addition to bisphosphonate treatment, supplementation with calcium and vitamin D may preserve bone after organ transplantation. Prior studies have compared bisphosphonates to calcium and vitamin D regimens. However, a combination regimen including each of these treatments may preserve bone mass better than a single treatment. Data regarding treatment with a combination of a bisphosphonate, calcium, and vitamin D are lacking in kidney and heart transplantation.

Comparison(s): In a prospective, open-label, single arm trial, Pamidronate (60-90 mg) is administered within 2 weeks after kidney or heart transplant and every 6 months for 2 years. Participants are prescribed vitamin D 800 units/d or calcitriol 0.25 microgram/d if serum creatinine is greater than 2 mg/dl, and calcium carbonate 1500 mg/d.

The primary outcome is bone mineral density measured by dual-energy X-ray absorptiometry at baseline and after years 1 and 2. Fracture events and serum calcium, parathyroid hormone, creatinine, and dipstick proteinuria are also measured.

ELIGIBILITY:
Inclusion Criteria:

* Kidney or heart transplant recipients

Exclusion Criteria:

* Hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 1999-01; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Bone mineral density measured by dual-energy X-ray absorptiometry | Every 12 months
  Performed at 1 year and 2 years.

SECONDARY OUTCOMES:
Fracture events | Every 6 months
  Evaluated at 6, 12, 18 months and 2 years
serum calcium | Every 6 months
  baseline, 6,12,18 months and 2 years
parathyroid hormone | Every 6 months
  baseline, 6,12,18 months and 2 years
serum creatinine and estimated glomerular filtration rate | Every 6 months
  Performed at 6,12,18 months and 2 years
proteinuria | Every 6 months
  Evaluated at 6,12,18 months and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R. Tuttle, MD,FASN,FACP, Principal Investigator — Providence Medical Research Center
Locations (1):
- Providence Medical Research Center, Spokane, Washington, United States